CLINICAL TRIAL: NCT05570227
Title: Identification of Metabolic Phenotypes Associated With Prognosis and Therapeutic Response in Patients With Melanoma
Brief Title: Metabolic Phenotypes in Melanoma
Acronym: MetaMel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21/164
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Melanoma
Keywords: Metabolism
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [U-13C]Glucose Infusion (Experimental): A 13.3% solution of sterile, pyrogen-free [U-13C]glucose in sterile water will be infused intravenously rapidly over 10 minutes to a total dose of 8 grams (bolus dose). Then the infusion will change to a rate of 4 grams/ hour. The infusion will continue until the time of tumour excision or biopsy, planned 2-3 hours.
  Interventions: Other: [U-13C]Glucose Infusion
- No [U-13C]Glucose Infusion (No Intervention): Blood and tissue samples to be collected for translational research studies, no other additional intervention.

INTERVENTIONS:
Other: [U-13C]Glucose Infusion — Peri-operative infusion of [U-13C]glucose
  Arms: [U-13C]Glucose Infusion

SUMMARY:
This is a single centre, correlative, longitudinal, biomarker study that aims to describe the metabolic features of human melanoma using mass spectrometry.

DETAILED DESCRIPTION:
This is a single-centre, correlative study designed to investigate metabolic phenotypes in a longitudinal cohort of patients with melanoma. This study will involve the collection of tissue at the time of surgical excision or biopsy. The key intervention, in a subset of patients, will be to perform peri-operative infusions of a stable isotope, [U13C]Glucose. Patients will be intravenously administered sterile, pyrogen-free 13C-glucose, delivered as an 8g bolus followed by infusion of 4g/hour for 2-3 hours. Blood samples will be obtained to monitor glucose and to analyse enrichment of labelled nutrients by gas-chromatography mass spectrometry (GC-MS). At the time of resection or biopsy, tumour samples will be divided and either immediately frozen in liquid nitrogen or processed to form patient-derived xenografts. Frozen tumour samples will be subsequently processed for: isotope enrichment by GC-MS; global metabolomics by liquid-chromatography mass spectrometry (LC-MS); and genomic analyses. Relevant clinical, histologic and genomic features will also be correlated with metabolic findings.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent
2. Male or female aged 18 years or older at written informed consent
3. Presence of a known melanoma lesion requiring surgical excision or biopsy
4. Patient is willing and able to comply with the protocol for the duration of the study including undergoing biopsies and receiving a stable isotope infusion (where applicable)

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from receiving a [U-13C]Glucose infusion:

1. Diabetes mellitus
2. Pregnancy or breast feeding
3. Patients unable to comply with study procedures and follow up in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Glucose Utilisation in the TCA cycle | 5 years
  In patients receiving a [U-13C]Glucose infusion, assess glucose utilisation in the TCA cycle (using the ratio of citrate M+2/pyruvate M+3, a surrogate of the pyruvate dehydrogenase reaction)
Lactate Utilisation in the TCA cycle | 5 years
  In patients receiving a [U-13C]Glucose infusion, assess lactate utilisation in the TCA cycle (using the ratio of lactate M+3/3PG M+3 as a surrogate measure)

SECONDARY OUTCOMES:
Relapse free survival | 5 years
  Defined as the time from surgery to disease recurrence or melanoma-related death, whichever occurs first
Overall Survival | 5 years
  Measured as the time of surgery until death from any cause

OTHER OUTCOMES:
Tumour Metabolomic and Lipidomic Profiling | 5 years
  Abundance of metabolites and lipid species, quantified by liquid chromatography mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Rao, MBBS PhD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter Mac Callum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No